CLINICAL TRIAL: NCT06117956
Title: Helicobacter Pylori in Patients With Chronic Tonsillits Prepared for Tonsillectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Fathy Abdelsattar, Resident- ENT DEPARTEMENT SUGAR COMPANY HOSPITAL, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: soh-Med-23-10-06 MS
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Infection in Patients With Chronic Tonsillits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid urease test for h pylori — Tonsillectomy will be done with the dissection method and one tonsil per patient will be collected. A 2 mm gross specimen will be washed with normal saline. The specimen will be placed in a test tube well containing Rapid Urease Enzyme (GASTRO CURE SYSTEM RUT DRY TEST Batch No. A1060).
  The initial color will be read at 0 min. Subsequent color changes will be read at 30 min, 6 hours, and 24 hours. Any color change from the initial yellow color to either pink or red will be recorded as positive. Any test that will be remained yellow after 24 hours will be recorded as negative.
  Tonsillar tissue samples will be fixed in 10% formalin for 24 h Each slide will be separately evaluated for the presence or absence of Helicobacter-like organisms at a high-power magnification
  Other Names: histopathological study for removed tonsillar tissue after tonsillectomy

SUMMARY:
Tonsillar disorders are frequent In both pediatric and adult otolaryngological practice, . Numerous disorders that damage tonsillar tissue necessitate tonsillectomy. Tonsillectomy is typically required for recurrent tonsillitis. (Mani et al., 2019).

According to studies, the mucosa-associated lymphoid tissue (MALT) of the stomach and tonsillar tissue in the Waldeyer's ring are both lymphoid tissues (Ma et al., 2018).

One of the most prevalent and frequent conditions in otorhinolaryngology is chronic tonsillitis, which is mostly brought on by bacterial infection. Chronic tonsillitis attacks can affect not only the tonsillar tissue but also can contribute to the emergence and progression of systemic disorders (Alrayah.,2023).

A gram-negative, urease-producing bacterium called Helicobacter pylori colonizes the mucosa of the digestive tract. It has been linked to gastric malignancies, notably mucosa-associated lymphoid tissue (MALT) lymphoma, as well as gastric ulcers and duodenal ulcers (Kusters et al., 2006).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 5 to 50 years.
2. Of both sex.
3. Diagnosed with chronic tonsillitis undergoing elective tonsillectomy

Exclusion Criteria:

1. Patients on proton pump inhibitor or antibiotics 2 weeks before surgery .
2. Immune-compromised patients.
3. Patients with obstructive sleep apnea candidates for adenotonsillectomy

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
positive or negative h pylori infection in tonsillar tissue after tonsillectomy | 6 months
  Tonsillectomy will be done with the dissection method and one tonsil per patient will be collected. A 2 mm gross specimen will be washed with normal saline. The specimen will be placed in a test tube well containing Rapid Urease Enzyme (GASTRO CURE SYSTEM RUT DRY TEST Batch No. A1060).
  The initial color will be read at 0 min. Subsequent color changes will be read at 30 min, 6 hours, and 24 hours. Any color change from the initial yellow color to either pink or red will be recorded as positive. Any test that will be remained yellow after 24 hours will be recorded as negative. No readings will be taken after 24 hours.
  Histopathology:
  Tonsillar tissue samples will be fixed in 10% formalin for 24 h. Each slide will be separately evaluated for the presence or absence of Helicobacter-like organisms at a high-power magnification

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt